CLINICAL TRIAL: NCT02468557
Title: A Phase 1b Study of Single Agent Idelalisib Followed by Idelalisib in Combination With Chemotherapy in Subjects With Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Study of Single Agent Idelalisib Followed by Idelalisib in Combination With Chemotherapy in Adults With Metastatic Pancreatic Ductal Adenocarcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-385-1577
Record Dates: First submitted 2015-06-08; First posted 2015-06-11 (Estimated); Results first posted 2021-03-22 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Previously Untreated Pancreatic Ductal Adenocarcinoma; Relapsed/Refractory Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Recurrence | interventions — idelalisib; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Idelalisib 150 mg (Experimental): Participants were administered with idelalisib (IDL) 150 mg tablets orally, twice daily (morning and evening) for 8 weeks.
  Interventions: Drug: Idelalisib
- Idelalisib + nab-paclitaxel (Experimental): Participants will receive escalating doses of idelalisib at a dose level of up to 150mg + nab-paclitaxel.
  Interventions: Drug: Idelalisib; Drug: Nab-paclitaxel
- Idelalisib + mFOLFOX6 (Experimental): Participants will receive escalating doses of idelalisib at a dose level of up to 150mg + mFOLFOX6.
  Interventions: Drug: Idelalisib; Drug: mFOLFOX6

INTERVENTIONS:
Drug: Idelalisib — Tablets administered orally twice daily
  Other Names: GS-1101; CAL-101; Zydelig®
Drug: Nab-paclitaxel — 125 mg/m^2 administered intravenously on Days 1, 8 and 15 of each 28 day cycle
  Arms: Idelalisib + nab-paclitaxel
Drug: mFOLFOX6 — mFOLFOX6 will be administered intravenously on Days 1 and 15 of each 28 day cycle. This regimen consists of levoleucovorin 200 milligram/meter per square (mg/m^2) or racemic leucovorin 400 mg/m^2, oxaliplatin 85 mg/m^2, bolus 5-fluorouracil 400 mg/m^2, and a 46 hour infusion of 5-fluorouracil 2, 400 mg/m^2.
  Arms: Idelalisib + mFOLFOX6

SUMMARY:
The primary objective of this study is to evaluate the safety of single agent idelalisib and to evaluate safety and define the maximum tolerated dose (MTD) of idelalisib in combination with chemotherapy in adults with metastatic pancreatic ductal adenocarcinoma.

ELIGIBILITY:
Key Inclusion Criteria:

* The presence of metastatic pancreatic adenocarcinoma plus 1 of the following:

  * Histological diagnosis of pancreatic adenocarcinoma confirmed pathologically, OR
  * Pathologist confirmed histological/cytological diagnosis of adenocarcinoma consistent with pancreas origin
* Measurable disease per response evaluation criteria in solid tumors (RECIST) v1.1
* Prior systemic chemotherapy treatment for metastatic pancreatic ductal adenocarcinoma (Arm: idelalisib single agent only)
* Received one prior line of chemotherapy for metastatic pancreatic ductal adenocarcinoma (Arm: idelalisib + mFOLFOX6 only)
* Adequate organ function defined as follows:

  * Hepatic: Total bilirubin ≤ 1.25 x upper limit of normal (ULN) (Arm: idelalisib + nab-paclitaxel ); total bilirubin ≤1.5 x ULN (Arm: single agent idelalisib and Arm: idelalisib + mFOLFOX6); aspartate transaminase (AST) serum glutamic oxaloacetic transaminase (SGOT), alanine transaminase (ALT) serum glutamic pyruvic transaminase (SGPT) < 2.5 x ULN, and albumin > 3.0 g/dL
  * Hematological: absolute neutrophil count (ANC) > 1,500 cells/cubic millimetre (m^3), platelet > 100,000 cells/mm^3, hemoglobin > 9.0 grams/decilitre (g/dL)
  * Renal: Serum creatinine ≤ 1.5 x ULN OR calculated creatinine clearance (CrCl) > 30 millilitre (ml)/min as calculated by the Cockcroft-Gault method
* Able to comprehend and willing to sign the written informed consent form

Key Exclusion Criteria:

* Currently or previously treated with biologic, or immunotherapy
* Currently or previously treated with conventional chemotherapy, or other agents for metastatic pancreatic ductal adenocarcinoma (Arm: idelalisib + nab-paclitaxel only)
* Evidence of ongoing systemic bacterial, fungal, or viral infection at the time of enrollment
* Known human immunodeficiency viruses (HIV) infection
* History of a concurrent or second malignancy except for adequately treated local basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy or requiring only hormonal therapy and with normal prostate-specific antigen for ≥ 1 year prior to enrollment, adequately treated Stage 1 or 2 non-pancreatic cancer currently in complete remission, or any other non-pancreatic cancer that has been in complete remission for ≥ 5 years
* Diagnosis of pancreatic islet neoplasm, acinar cell carcinoma, non-adenocarcinoma (eg, lymphoma, sarcoma), adenocarcinoma originating from the biliary tree or cystadenocarcinoma
* History of serious allergic reaction, including anaphylaxis and toxic epidermal necrolysis
* Presence of peripheral neuropathy ≥ Grade 2 (Arm: idelalisib + nab-paclitaxel and Arm: idelalisib + mFOLFOX6)
* Documented myocardial infarction or unstable/uncontrolled cardiac disease (eg, unstable angina, congestive heart failure [New York Heart Association > Class III]) within 6 months or enrollment
* Known hypersensitivity to idelalisib, its metabolites, or formulation excipients
* Known hypersensitivity to nab-paclitaxel (Arm: idelalisib + nab-paclitaxel), their metabolites, or formulation excipients
* Known hypersensitivity to 5-fluorouracil, leucovorin, or oxaliplatin (Arm: idelalisib + mFOLFOX6), their metabolites, or formulation excipients

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-07-30 (Actual); Primary Completion 2016-04-27 (Actual); Study Completion 2016-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (9):
- United States (9):
  - Scottsdale Healthcare Clinical Research Institute, Scottsdale, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - Indiana University Goshen Center for Cancer Care, Goshen, Indiana
  - Dana Farber/ Harvard Cancer Institute, Boston, Massachusetts
  - University of Rochester, Rochester, New York
  - Greenville Hospital System, Greenville, South Carolina
  - Mary Crowley Medical Research Center, Dallas, Texas

REFERENCES:
- [Background] Borazanci E, Pishvaian MJ, Nemunaitis J, Weekes C, Huang J, Rajakumaraswamy N. A Phase Ib Study of Single-Agent Idelalisib Followed by Idelalisib in Combination with Chemotherapy in Patients with Metastatic Pancreatic Ductal Adenocarcinoma. Oncologist. 2020 Nov;25(11):e1604-e1613. doi: 10.1634/theoncologist.2020-0321. Epub 2020 Jun 18. PMID 32356383

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 30 July 2015. The last study visit occurred on 27 April 2016.
Pre-assignment Details: 35 participants were screened. The study was terminated. No participants were enrolled in the Idelalisib (IDL) + nab-paclitaxel or IDL + mFOLFOX [5- fluorouracil (FU), leucovorin and oxaliplatin] groups.
Period: Overall Study
Arm/Group | Idelalisib 150 mg
Started | 16
Completed | 0
Not Completed | 16
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Study Terminated by Sponsor, Regulatory Agency or Institutional Review Board/ Ethics Committee | 10
Not completed — All Enrolled but Never Dosed | 4

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set included all participants who received at least 1 dose of study drug.
Arm/Group | Idelalisib 150 mg
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted means local regulators did not allow collection of race information.
  Participants
    Race: American Indian or Alaska Native | 0
    Race: Asian | 0
    Race: Black | 1
    Race: Native Hawaiian or Pacific Islander | 0
    Race: White | 11
    Race: Other | 0
    Race: Not Permitted | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted means local regulators did not allow collection of ethnicity information.
  Participants
    Ethnicity: Hispanic or Latino | 0
    Ethnicity: Not Hispanic or Latino | 12
    Ethnicity: Not Permitted | 0

OUTCOME MEASURES:

1. Primary Outcome: Single-agent IDL: Percentage of Participants Who Experienced Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as adverse events (AEs) with onset dates on or after the study drug start date and no later than 30 days after the permanent discontinuation of the study drug. It also included the AEs that led to premature discontinuation of study drug.
Time Frame: First dose date up to last dose date (Maximum: 8 weeks) plus 30 days
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Idelalisib 150 mg
Number analyzed (Participants) | 12
percentage of participants | 100.0

2. Primary Outcome: Single-agent IDL: Percentage of Participants Who Experienced Treatment-Emergent Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increased at least 1 toxicity grade from baseline at any post baseline time point, up to and including the date of last dose of study drug plus 30 days. If the relevant baseline laboratory value was missing, any abnormality of at least Grade 1 observed within the time frame specified above was considered treatment emergent. Severity grade is defined by Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 (1=Mild, 2=Moderate, 3=Severe, 4=Life-threatening). The percentage of participants for any post-baseline abnormal laboratory value in the Grade 1-4 category is reported. The term 'hypo' indicates less than the normal count of a parameter and 'hyper' indicates more than the normal count of a parameter.
Time Frame: First dose date up to last dose date (Maximum: 8 weeks) plus 30 days
Population: Participants in the safety analysis set were analysed.
Measure: Number; unit: percentage of participants
Arm/Group | Idelalisib 150 mg
Number analyzed (Participants) | 12
percentage of participants
  Hemoglobin (Hypo), Hematology | 25.0
  Lymphocytes (Hyper), Hematology | 8.3
  Lymphocytes (Hypo), Hematology | 25.0
  Platelets, Hematology | 8.3
  Alanine Aminotransferase, Chemistry | 58.3
  Albumin, Chemistry | 16.7
  Alkaline Phosphatase, Chemistry | 33.3
  Aspartate Aminotransferase, Chemistry | 66.7
  Bilirubin, Chemistry | 16.7
  Creatinine Clearance, Chemistry | 16.7
  Gamma Glutamyl Transferase, Chemistry | 50.0
  Glucose (Hyper), Chemistry | 16.7
  Sodium (Hypo), Chemistry | 25.0

3. Primary Outcome: Idelalisib in Combination With Chemotherapy: Percentage of Participants With Dose Limiting Toxicities (DLTs)
Description: Dose limiting toxicities were defined as toxicities experienced during the first 28 days of treatment (Cycle 1) that were judged to be clinically significant and at least possibly related to study treatment.
Time Frame: Up to 28 days
Population: Due to the early termination of the study, there were no participants enrolled in the Idelalisib Combination arms.
Groups:
- Idelalisib + Nab-paclitaxel: Participants were to be administered IDL tablets orally twice daily plus nab-paclitaxel administered intravenously on Days 1, 8 and 15 of each 28 day cycle.
- Idelalisib + mFOLFOX6: Participants were to be administered IDL tablets orally twice daily plus mFOLFOX6 administered intravenously on Days 1 and 15 of each 28 day cycle.
Arm/Group | Idelalisib + Nab-paclitaxel | Idelalisib + mFOLFOX6
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in FoxP3+ and Cluster Determinant 8+ (CD8+) Cells From Tumor Tissue Samples as a Measure of Pharmacodynamics Activity
Time Frame: Up to 2 years
Population: Due to the early termination of the study no pharmacodynamic testing was performed.
Arm/Group | Idelalisib 150 mg | Idelalisib + Nab-paclitaxel | Idelalisib + mFOLFOX6
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Idelalisib Plasma Concentrations Following Idelalisib 150 mg Twice Daily
Time Frame: Cycle 1, Day 1: Predose and 0.5, 1, 1.5, 2, 3, 4, and 8 hours (h) postdose; Day 8: Predose and 1.5 h postdose; Day 15: Predose and 1.5 h postdose Cycle 2, Day 1: Predose and 1.5 h postdose
Population: The pharmacokinetic (PK) Analysis Set included all participants in the Full Analysis Set who had the necessary baseline and on-study measurements to provide interpretable results for the specific parameters of interest. Due to the early termination of the study, concentration data is reported because there was an insufficient number of participants sampled for PK analysis to generate PK parameters.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Idelalisib 150 mg
Number analyzed (Participants) | 12
ng/mL
  Cycle 1; Day 1 (Predose): number analyzed (Participants) | 7
  Cycle 1; Day 1 (Predose) | NA [NA to NA] — The plasma concentration of IDL was below the limit of quantitation.
  Cycle 1; Day 1 (0.5 h): number analyzed (Participants) | 3
  Cycle 1; Day 1 (0.5 h) | 1110 [13.90 to 3220]
  Cycle 1; Day 1 (1 h): number analyzed (Participants) | 3
  Cycle 1; Day 1 (1 h) | 1880 [39.10 to 4060]
  Cycle 1; Day 1 (1.5 h): number analyzed (Participants) | 11
  Cycle 1; Day 1 (1.5 h) | 1690 [318 to 2260]
  Cycle 1; Day 1 (2 h): number analyzed (Participants) | 3
  Cycle 1; Day 1 (2 h) | 1290 [173 to 4460]
  Cycle 1; Day 1 (3 h): number analyzed (Participants) | 3
  Cycle 1; Day 1 (3 h) | 795 [631 to 2870]
  Cycle 1; Day 1 (4 h): number analyzed (Participants) | 3
  Cycle 1; Day 1 (4 h) | 1540 [519 to 1990]
  Cycle 1; Day 1 (8 h): number analyzed (Participants) | 3
  Cycle 1; Day 1 (8 h) | 251 [134 to 753]
  Cycle 1; Day 8 (Predose): number analyzed (Participants) | 8
  Cycle 1; Day 8 (Predose) | 264 [208 to 501.5]
  Cycle 1; Day 8 (1.5 h): number analyzed (Participants) | 8
  Cycle 1; Day 8 (1.5 h) | 2050 [1335 to 2620]
  Cycle 1; Day 15 (Predose): number analyzed (Participants) | 3
  Cycle 1; Day 15 (Predose) | 275 [241 to 1120]
  Cycle 1; Day 15 (1.5 h): number analyzed (Participants) | 4
  Cycle 1; Day 15 (1.5 h) | 1605 [1170 to 2130]
  Cycle 2; Day 1 (Predose): number analyzed (Participants) | 4
  Cycle 2; Day 1 (Predose) | 178.05 [39.05 to 281]
  Cycle 2; Day 1 (1.5 h): number analyzed (Participants) | 4
  Cycle 2; Day 1 (1.5 h) | 2180 [1825 to 3095]

6. Secondary Outcome: Idelalisib Metabolite (GS-563117) Plasma Concentrations Following Idelalisib 150 mg Twice Daily
Time Frame: Cycle 1, Day 1: Predose and 0.5, 1, 1.5, 2, 3, 4, and 8 h postdose; Day 8: Predose and 1.5 h postdose; Day 15: Predose and 1.5 h postdose Cycle 2, Day 1: Predose and 1.5 h postdose
Population: Participants in the PK Analysis Set with available data were analysed. Due to the early termination of the study, concentration data is reported because there was an insufficient number of participants sampled for PK analysis to generate PK parameters.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Idelalisib 150 mg
Number analyzed (Participants) | 12
ng/mL
  Cycle 1; Day 1 (Predose): number analyzed (Participants) | 7
  Cycle 1; Day 1 (Predose) | NA [NA to NA] — The plasma concentration of GS-563117 was below the limit of quantitation.
  Cycle 1; Day 1 (0.5 h): number analyzed (Participants) | 3
  Cycle 1; Day 1 (0.5 h) | 173 [NA to 220] — The plasma concentration of GS-563117 was below the limit of quantitation.
  Cycle 1; Day 1 (1 h): number analyzed (Participants) | 3
  Cycle 1; Day 1 (1 h) | 1220 [16.70 to 1460]
  Cycle 1; Day 1 (1.5 h): number analyzed (Participants) | 11
  Cycle 1; Day 1 (1.5 h) | 1070 [141 to 1930]
  Cycle 1; Day 1 (2 h): number analyzed (Participants) | 3
  Cycle 1; Day 1 (2 h) | 1700 [106 to 4430]
  Cycle 1; Day 1 (3 h): number analyzed (Participants) | 3
  Cycle 1; Day 1 (3 h) | 1580 [190 to 5980]
  Cycle 1; Day 1 (4 h): number analyzed (Participants) | 3
  Cycle 1; Day 1 (4 h) | 1370 [849 to 5960]
  Cycle 1; Day 1 (8 h): number analyzed (Participants) | 3
  Cycle 1; Day 1 (8 h) | 632 [619 to 5340]
  Cycle 1; Day 8 (Predose): number analyzed (Participants) | 8
  Cycle 1; Day 8 (Predose) | 2175 [1385 to 5790]
  Cycle 1; Day 8 (1.5 h): number analyzed (Participants) | 8
  Cycle 1; Day 8 (1.5 h) | 2775 [1765 to 5725]
  Cycle 1; Day 15 (Predose): number analyzed (Participants) | 3
  Cycle 1; Day 15 (Predose) | 2130 [1020 to 6800]
  Cycle 1; Day 15 (1.5 h): number analyzed (Participants) | 4
  Cycle 1; Day 15 (1.5 h) | 2890 [2010 to 4815]
  Cycle 2; Day 1 (Predose): number analyzed (Participants) | 4
  Cycle 2; Day 1 (Predose) | 1046.5 [490.34 to 1360]
  Cycle 2; Day 1 (1.5 h): number analyzed (Participants) | 4
  Cycle 2; Day 1 (1.5 h) | 1405 [1325 to 2305]

7. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response rate (ORR) was defined as the percentage of participants who achieved a Complete Response (CR) or Partial Response (PR) as assessed by response evaluation criteria in sold tumors (RECIST) v1.1.
Time Frame: Up to 2 years
Population: Due to early study termination, the prespecified efficacy analyses were not conducted.
Arm/Group | Idelalisib 150 mg | Idelalisib + Nab-paclitaxel | Idelalisib + mFOLFOX6
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the interval from first dose date of study drug to death from any cause.
Time Frame: Up to 2 years
Population: Due to early study termination, the prespecified efficacy analyses were not conducted.
Arm/Group | Idelalisib 150 mg | Idelalisib + Nab-paclitaxel | Idelalisib + mFOLFOX6
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival is defined as the interval from first dose date of study drug to the earlier of the first documentation of definitive disease progression or death from any cause.
Time Frame: Up to 2 years
Population: Due to early study termination, the prespecified efficacy analyses were not conducted.
Arm/Group | Idelalisib 150 mg | Idelalisib + Nab-paclitaxel | Idelalisib + mFOLFOX6
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to last dose date (Maximum: 8 weeks) plus 30 days All-cause mortality: First dose date up to study termination (approximately 39 weeks)
Description: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Arm/Group | Idelalisib 150 mg
All-Cause Mortality (participants affected / at risk) | 2/12
Serious Adverse Events (participants affected / at risk) | 3/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib 150 mg (N=12)
Coagulopathy (Blood and lymphatic system disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib 150 mg (N=12)
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Rectal spasm (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Chills (General disorders) | 2
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 5
Xerosis (General disorders) | 1
Bacteraemia (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 4
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Weight decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Aphasia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 2
Chromaturia (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Urinary tract obstruction (Renal and urinary disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Rash macular (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Due to the early termination of the study, the prespecified efficacy, pharmacodynamic, and pharmacokinetic analysis for PK parameters were not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years